CLINICAL TRIAL: NCT03382457
Title: Clinical Study of Edwards Cardioband FIT Valve Repair System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-19
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Tricuspid Regurgitation
Keywords: Functional; TR; FTR; Transcatheter; Repair
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Treatment with the Edwards Cardioband FIT Repair System
  Interventions: Device: Transcatheter Tricuspid Valve Repair

INTERVENTIONS:
Device: Transcatheter Tricuspid Valve Repair — Repair of the tricuspid valve through a transcatheter approach
  Other Names: Edwards Cardioband Tricuspid Valve Repair

SUMMARY:
Clinical Study of the Edwards Cardioband FIT Repair System

DETAILED DESCRIPTION:
The study is a multi-center, prospective, single-arm, and non-randomized study designed to evaluate the safety and performance of the Edwards Cardioband FIT Repair System

ELIGIBILITY:
Key Inclusion Criteria:

* Tricuspid regurgitation (moderate or greater)
* Despite medical therapy, per the local Heart Team, patient has signs of TR, symptoms from TR, or prior heart failure hospitalization from TR.
* The local site Heart Team determines that the patient is appropriate for transcatheter tricuspid reconstruction
* Patient is willing and able to comply with all specified study evaluations and provides written informed consent

Key Exclusion Criteria:

Patients with conditions or anatomical considerations that preclude safe and successful procedure-related or study device access, deployment, or function, including but not limited to:

* Patients in whom transesophageal echocardiography is contraindicated or cannot be completed.
* Patients in whom tricuspid valve anatomy is not evaluable by TTE or TEE
* Untreatable hypersensitivity or contraindication to any of the following: all antiplatelets, all anticoagulants, nitinol alloys (nickel and titanium), polyester, or contrast media.
* Previous tricuspid valve repair or replacement with device in place
* Presence of trans-tricuspid pacemaker or defibrillator leads where: (a)TR is a result of impingement on the tricuspid valve leaflet as evaluated by echocardiography; or (b) implanted in the RV within the last 90 days

Primary tricuspid valve disease

Any physical impairment which limits the patient's capacity to complete functional testing due to other medical conditions independent of their TR (e.g., orthopedic condition)

Currently participating in another investigational biologic, drug, or device study

Any of the following cardiovascular procedures:

* Percutaneous coronary, intracardiac, or endovascular intervention within the last 30 days
* Carotid surgery within the last 30 days
* Direct current cardioversion within the last 30 days
* Leadless RV pacemaker implant within the last 30 days
* Cardiac surgery within the last 90 days

Any of the following underlying medical conditions:

* Severe aortic, mitral and/or pulmonic valve stenosis and/or regurgitation
* Active endocarditis or infection requiring antibiotic therapy (oral or intravenous)
* Hemodynamically significant pericardial effusion
* Significant intra-cardiac mass, thrombus, or vegetation
* Untreated clinically significant coronary artery disease (CAD) requiring revascularization, evidence of acute coronary syndrome, or recent myocardial infarction (MI)
* Known history of untreated severe symptomatic carotid stenosis (>50% by ultrasound) or asymptomatic carotid stenosis (>70% by ultrasound)
* Hypotension (systolic pressure <90 mmHg) or requirement for inotropic support or hemodynamic support within the last 30 days
* Known bleeding or clotting disorders or patient refuses blood transfusion
* Active GI bleeding
* Recent stroke
* Need for emergent or urgent surgery for any reason or any planned cardiac surgery within the next 12 months or any planned percutaneous cardiac procedure within the next 90 days
* Deep vein thrombosis (DVT) or pulmonary embolism (PE) in the last 6 months

Pregnant, breastfeeding, or planning pregnancy within the next 12 months

Concurrent medical condition with a life expectancy of less than 12 months in the judgment of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint -Composite Major Adverse Event (MAE) Rate | 30 days
  Number and percentage of patients who experienced at least one major adverse event (MAE).
Primary Performance Endpoint - Intraprocedural Success | Intraprocedural
  Number of patients who had Intraprocedural Success, definition modified from TVARC criteria. Per patient analysis.
Primary Performance Endpoint - Clinical Success | 30 days and 1 year
  Number of patients who had Clinical Success at 30 days and 1 year, definition modified from TVARC criteria. Per patient analysis.

CONTACTS AND LOCATIONS:
Overall Officials: William Gray, MD, Principal Investigator — Lankenau Heart; Firas Zahr, MD, Principal Investigator — Oregon Health and Science University
Locations (9):
- United States (9):
  - Northwestern University, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Morristown Medical Center, Morristown, New Jersey
  - Columbia University Medical Center /New York Presbyterian Hospital, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Heart Hospital Baylor Plano, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davidson CJ, Abramson S, Smith RL, Kodali SK, Kipperman RM, Eleid MF, Reisman M, Whisenant BK, Puthumana J, Fowler D, Grayburn PA, Hahn RT, Koulogiannis K, Pislaru SV, Zwink T, Minder M, Deuschl F, Feldman T, Gray WA, Lim DS; Cardioband Tricuspid Valve Reconstruction System Early Feasibility Study Investigators. Transcatheter Tricuspid Repair With the Use of 4-Dimensional Intracardiac Echocardiography. JACC Cardiovasc Imaging. 2022 Mar;15(3):533-538. doi: 10.1016/j.jcmg.2021.01.029. Epub 2021 Mar 17. No abstract available. PMID 33744150
- [Derived] Davidson CJ, Lim DS, Smith RL, Kodali SK, Kipperman RM, Eleid MF, Reisman M, Whisenant B, Puthumana J, Abramson S, Fowler D, Grayburn P, Hahn RT, Koulogiannis K, Pislaru SV, Zwink T, Minder M, Dahou A, Deo SH, Vandrangi P, Deuschl F, Feldman TE, Gray WA; Cardioband TR EFS Investigators. Early Feasibility Study of Cardioband Tricuspid System for Functional Tricuspid Regurgitation: 30-Day Outcomes. JACC Cardiovasc Interv. 2021 Jan 11;14(1):41-50. doi: 10.1016/j.jcin.2020.10.017. PMID 33413863